CLINICAL TRIAL: NCT06296589
Title: Clinical Effectiveness and Implementation of Trauma-Informed Guilt Reduction Therapy Compared to Prolonged Exposure (TrIGR)
Brief Title: Trauma-Informed Guilt Reduction Therapy Compared to Prolonged Exposure
Acronym: PORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: University of Minnesota (Other); Center for Veterans Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HT94252310861
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trauma Informed Guilt Reduction Therapy (Experimental): 6 session behavioral intervention focused on trauma-related guilt, shame, and moral injury
  Interventions: Behavioral: Trauma Informed Guilt Reduction Therapy
- Prolonged Exposure Therapy (Active Comparator): 12 session behavioral intervention focused on PTSD symptoms
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Trauma Informed Guilt Reduction Therapy — Behavioral therapy for trauma related guilt and shame
  Arms: trauma Informed Guilt Reduction Therapy
Behavioral: Prolonged Exposure Therapy — Behavioral exposure therapy for PTSD
  Arms: Prolonged Exposure Therapy

SUMMARY:
The goal of this clinical trial is to learn if receiving Trauma-Informed Guilt Reduction (TrIGR) Therapy is as effective as receiving Prolonged Exposure Therapy among veterans with PTSD and trauma related guilt. The main questions it aims to answer are:

Will TrIGR be comparable to PE in terms of PTSD symptom reduction? Will it TrIGR be comparable to PE in improving functioning and reducing depression symptoms? Will it be superior in improving trauma-related guilt and shame?

DETAILED DESCRIPTION:
Trauma-related guilt is common and impairing among trauma survivors. Guilt is positively associated with severity of PTSD and depression symptoms, poorer psychosocial functioning and suicide risk. Although existing evidence-based trauma-focused PTSD treatments such as Prolonged Exposure (PE) are effective in treating PTSD and trauma-related guilt, many still experience symptoms or maintain their diagnosis after treatment. Preliminary research shows that a brief treatment targeting trauma-related and moral injury-related guilt and shame, Trauma Informed Guilt Reduction Therapy (TrIGR), can reduce guilt, PTSD, depression, and distress among Veterans and help them reengage with meaningful activities. Whether TrIGR is comparably effective to longer, more resource heavy evidence-based PTSD treatments disseminated across DoD and VA, like PE, is a critical question.

The proposed randomized clinical trial aims to determine if TrIGR is non-inferior to a first tier PTSD treatment, PE. Hypotheses are that 6 sessions of TrIGR will be non-inferior to 12 sessions of PE in reducing PTSD symptom severity among Veterans with PTSD who endorse trauma-related guilt. Secondary aims are to evaluate the hypotheses that TrIGR will be non-inferiority relative to PE in improving psychosocial functioning and depression symptoms and superior in reducing trauma-related guilt and shame. The study will also explore treatment differences in change in suicidal ideation and dropout.

Participants will be recruited from mental health clinics across three VAs. 158 Veterans who served since 9/11 and with PTSD and guilt from any type of trauma will be included. TrIGR will be administered over 6 weekly sessions (60-minutes each) and PE will be administered over 12 weekly sessions (90 minutes each). Blind assessors will evaluate participants at baseline and 8-, 16-, and 28 weeks after the first therapy session. Inclusion and exclusion criteria are minimized so that generalizability will be high.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veterans age 18 or older who served in the military since the start of Operation Enduring Freedom/Operation Iraqi Freedom; OEF/OIF)
* meets diagnostic criteria for PTSD;
* a score of 2 or higher ("true" to "extremely true") on feeling trauma-related guilt much or all of the time or scoring 3 or higher ("very true" or "extremely true") on at least one guilt cognition factor (hindsight bias/responsibility, wrongdoing, or lack of justification) on the Trauma Related Guilt Inventory
* not currently receiving trauma-focused treatment such as PE or CPT
* willingness to attend psychotherapy and assessment sessions

Exclusion Criteria:

* current risk of suicidal/homicidal behavior that requires immediate intervention
* current severe substance use disorder (in the past two months) based on DSM-5 criteria
* current unmanaged psychosis or mania
* life threatening or unstable medical illness
* inability to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 158 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | baseline and 8-, 16-, and 28 weeks after the first therapy session
  Measures PTSD symptom severity, score range 0-80, higher scores mean greater symptom severity

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | baseline and 8-, 16-, and 28 weeks after the first therapy session
  Depression symptom severity, range = 0-27, higher scores mean greater depression symptom severity
Brief Psychosocial Functioning Inventory (B-IPF) | baseline and 8-, 16-, and 28 weeks after the first therapy session
  Measures severity of impairment in psychosocial functioning, scores = 0-100, higher scores indicate greater impairment
Trauma Related Guilt Inventory Cognitions Scale (TRGI) | baseline and 8-, 16-, and 28 weeks after the first therapy session
  Measures severity of trauma related guilt cognitions, scores = 0-4, higher scores indicate greater guilt
Trauma Related Shame Inventory (TRSI) | baseline and 8-, 16-, and 28 weeks after the first therapy session
  Measures severity of trauma related shame, scores = 0-96, higher scores indicate greater shame

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Kehle-Forbes, PhD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Little Rock Veterans Health Care System (LRVHCS), Little Rock, Arkansas
  - Southeast Louisiana Veterans Health Care System (SLVHCS), New Orleans, Louisiana
  - William S. Middleton Memorial Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Will share data with Strong Star Repository.
Supporting Information: Study Protocol
Time Frame: After study completion.
Access Criteria: Request to StrongStar Repository that Strong Star must approve.
URL: http://www.strongstar.org/research/strongstar/strong-star-repository